CLINICAL TRIAL: NCT00026520
Title: Evaluation of Interferon Alpha-2b and Thalidomide in Patients With Disseminated Malignant Melanoma, Phase II
Brief Title: Interferon Alfa and Thalidomide in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069046; SWOG-S0026
Record Dates: First submitted 2001-11-09; First posted 2003-06-25 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2003-04

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Interferon-alpha; Thalidomide

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: thalidomide

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells and slow the growth of the tumor. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. Combining interferon alfa with thalidomide may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining interferon alfa with thalidomide in treating patients who have stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 6-month progression-free survival rate in patients with stage IV melanoma treated with interferon alfa and thalidomide.
* Determine the confirmed and unconfirmed complete and partial response rates in patients with measurable disease treated with this regimen.
* Determine the quantitative and qualitative toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive interferon alfa subcutaneously twice daily and oral thalidomide once daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) receive 2 additional courses after documentation of CR.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV malignant melanoma

  * Surgically incurable disease
* Measurable or evaluable disease
* No brain metastases by CT scan or MRI

  * Prior brain metastases allowed only if completely resected and treated with whole brain radiotherapy
* Must have received 1, and only 1, prior systemic therapy for metastatic disease

  * Chemotherapy, biologic/immunotherapy, hormonal therapy, or combination therapy

PATIENT CHARACTERISTICS:

Age:

* Adult

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3

Hepatic:

* SGOT and/or SGPT no greater than 2.5 times upper limit of normal (ULN)
* Bilirubin no greater than ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 methods of effective contraception 4 weeks before, during, and for 4 weeks after study
* HIV negative
* No AIDS or HIV-1-associated complex
* No other serious illness
* No serious active infections
* No sensory neuropathy greater than grade 1
* No prior seizures or concurrent potential risk factors for the development of seizures
* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 21 days since prior biologic therapy or immunotherapy in the adjuvant or metastatic setting and recovered
* No concurrent filgrastim (G-CSF)
* No other concurrent biologic therapy

Chemotherapy:

* See Disease Characteristics
* At least 21 days since prior chemotherapy in the adjuvant or metastatic setting and recovered
* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* At least 21 days since prior hormonal therapy in the adjuvant or metastatic setting and recovered
* No concurrent hormonal therapy
* No concurrent systemic steroids (including creams)

Radiotherapy:

* See Disease Characteristics
* At least 21 days since prior radiotherapy and recovered
* Prior radiotherapy to all known sites of disease allowed if there is objective evidence of progression
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 21 days since prior surgery for primary or metastatic disease and recovered
* No concurrent surgery

Other:

* At least 21 days since prior systemic therapy or combination regimen for metastatic disease and recovered
* At least 21 days since prior adjuvant isolation limb perfusion therapy and recovered
* No other concurrent therapy
* No other concurrent investigational drugs
* No concurrent immunosuppressive medications
* Concurrent antihistamines allowed if no alternative medication available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-11; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura F. Hutchins, MD, Study Chair — University of Arkansas
Locations (94):
- United States (94):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Result] Hutchins LF, Moon J, Clark JI, Thompson JA, Lange MK, Flaherty LE, Sondak VK. Evaluation of interferon alpha-2B and thalidomide in patients with disseminated malignant melanoma, phase 2, SWOG 0026. Cancer. 2007 Nov 15;110(10):2269-75. doi: 10.1002/cncr.23035. PMID 17932881
- [Result] Hutchins L, Moon J, Clark J, et al.: Interferon alpha-2b and thalidomide in previously treated patients with disseminated malignant melanoma: SWOG 0026. [Abstract] J Clin Oncol 22 (Suppl 14): A-7527, 716s, 2004.